CLINICAL TRIAL: NCT06180382
Title: Comparison of Vedolizumab Treatment to Adalimumab Dose Intensification in Crohn's Disease Patients With Loss of Response or Biomarker Activity to Adalimumab on First Line With Therapeutic Drug Concentration: A Randomized, Multicentre, Controlled Trial
Brief Title: Comparison of Vedolizumab Treatment to Adalimumab Dose Intensification in Crohn's Disease Patients With Loss of Response or Biomarker Activity to Adalimumab on First Line With Therapeutic Drug Concentration.
Acronym: VEDIAN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Takeda France (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23CH214; 2023-508154-25-00 (Other: CTIS)
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; Adalimumab; Vedolizumab; therapeutic strategy; Efficacy; biomarker
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab; vedolizumab

STUDY DESIGN:
Intervention Model Description: Randomization comparing 2 therapeutic strategies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adalimumab with optimisation (Experimental): Patients with Crohn's disease will be included. They will have Adalimumab with optimisation as treatment.
  Interventions: Drug: Adalimumab
- Vedolizumab (Experimental): Patients with Crohn's disease will be included. They will have Vedolizumab as treatment.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Adalimumab — Administration of adalimumab with optimisation either 80 mg every 14 days by subcutaneous injection, or the same dose of 40 mg every 7 days.
  Arms: Adalimumab with optimisation
Drug: Vedolizumab — Strategy B: administration of vedolizumab 300mg by infusion at baseline, 14 days, 42 days and 60 days, followed by a dose of 108mg every fortnight by subcutaneous injection.
  Arms: Vedolizumab

SUMMARY:
A substantial fraction of IBD patients with an initial response to infliximab or adalimumab later experience re-emerging active disease despite ongoing anti-Tumour Necrosis Factor (TNF) agents maintenance therapy. The optimal intervention in patients with secondary loss-of-response (LOR) is still poorly defined, as there are still scant data on how best to choose the next intervention from among dose-intensification, switch to another anti-TNF or switch out of the anti-TNF class. Moreover, according to STRIDE 2 recommendations and CALM study, optimize patients based solely on lack of biological remission (CRP, calprotectin) can be discuss. If CALM study has showed that the intervention arm based on regular monitoring fecal calprotectin, CRP and/or CDAI to optimize patients under adalimumab was significantly associated to an increase rate of mucosal healing that the standard of care strategy based on only clinical activity, TDM was not available to guide drug optimization strategy.

DETAILED DESCRIPTION:
To address these issues, for IFX or ADA therapy, several studies have proposed some algorithms according to which interventions are based on a combined assessment of IFX or ADA drug level and antibodies-to-IFX or ADA (ATI or AAA) levels at the time of therapeutic failure. Thus, IFX or ADA levels, classified as therapeutic or sub-therapeutic, and detectable or undetectable antibodies, are used to assess if LOR is likely due to immunogenicity, to non-immune-mediated pharmacokinetic problems or due to pharmacodynamic issues, and to guide interventions accordingly.

In the last AGA recommendations, the authors suggested that in case of secondary LOR under anti TNF drug with therapeutic levels to switch to another class (such as vedolizumab). However, recent studies showed that optimization of dose regimen of the same anti-TNF in these patients may still be associated with clinical response in 25% of patients. Indeed, in a recent bicentric, retrospective and non-randomized study, the investigators showed that IBD patients under ADA maintenance therapy who experience a secondary loss of response and in whom trough levels are >4.9µg/mL, swapping to another class was significantly better than optimizing ADA, in term of time without discontinuation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Major patient and having given consent to participate in the study
* Patients with Crohn's disease who have responded primary to Adalimumab princeps or similar bio with loss of response to Adalimumab (40 mg every two weeks) with therapeutically adequate levels of ADA (> 7.5 μg/mL).
* Patient affiliated to or entitled under a social security scheme

Exclusion Criteria:

* Pregnant woman
* Patient unable to perform MRI or VCE or ileocolonoscopy or ultrasound less than one month before inclusion
* Previous or current use of vedolizumab or ustekinumab for Crohn's disease or participation in a biological study
* Concomitant use of immunomodulators
* Patients on corticosteroid therapy
* History of cancer
* History of human immunodeficiency virus (HIV), immunodeficiency syndrome, central nervous system (CNS) demyelinating disease (including myelitis), neurological symptoms suggestive of demyelinating disease, chronic recurrent infection, active tuberculosis (received or untreated), severe infections such as sepsis and opportunistic infections
* Patient with ileoanal pouchitis or ileorectal anastomosis
* Patient with short small bowel syndrome as determined by investigator
* Patients receiving total parenteral nutrition (TPN)
* Patients receiving enteral nutrition
* Patient under legal protection or unable to give consent
* Hemorrhagic rectocolitis or indeterminate colitis
* Patients treated with concomitant immunosuppressive agents
* Patient treated with an optimized dose of adalimumab
* Primary non-responder to Adalimumab
* Patient previously treated with infliximab or ustekinumab before adalimumab
* Severe relapse defined by CDAI > 330
* Patient with anoperineal Crohn's disease
* Crohn's disease patient with transient or permanent stoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
ADA optimized versus Vedolizumab as second line | Week 24
  The primary objective will be to compare the proportion of clinical and biomarker remission (composite score) in the two groups of CD patients by 24 weeks after inclusion.

SECONDARY OUTCOMES:
Proportion of deep remission | Weeks 0; 24
  To compare the proportion of deep remissions, the composite score is :
  * Clinical and biomarker remission at week 24 ;
  * AND Mucosal remission at week 24;
  * AND no treatment failure between inclusion and week 24.
Proportion of clinical remission | Weeks 0; 24
  A patient is considered to be in clinical remission if they present:
  * A Crohn's Disease Activity Index (CDAI score) < 150 at week 24 ;
  * OR a CDAI score ≥ 150 at week 24 AND a CDAI score < 150 at inclusion AND an increase < 70 points between inclusion and week 24.
  CDAI is the Crohn's disease activity score most commonly used in clinical trials. A CDAI below 150 corresponds to inactive Crohn's disease; between 150 and 450 to active Crohn's disease; above 450 to severe Crohn's disease.
faecal calprotectin (microG / g) | Week 24
  Biomarkers are considered to be standardised if the following are observed
  - normalisation of faecal calprotectin: faecal calprotectin < 250 µg/g at week 24.
serum C-reactive protein (CRP) mg/l | Week 24
  Biomarkers are considered to be standardised if the following are observed
  - Normalisation of serum C-reactive protein (CRP) : serum CRP < 5 mg/L at week 24 ;
Proportion of endoscopic remissions according to Crohn's Disease Endoscopic Index score (CDEIS) | Week 24
  A patient is considered to be in endoscopic remission if they have:
  - a CDEIS score < 3 at week 24 using ileocolonoscopy ; The CDEIS is an index of the severity of intestinal lesions caused by Crohn's disease.
  The CDEIS ranges from 0 to 44 0: no lesions 44: most severe lesions Endoscopic remission defined by a CDEIS ≤ 7
Proportion of endoscopic remissions according to Lewis score | Week 24
  A patient is considered to be in endoscopic remission if they have:
  - a Lewis score < 135 at week 24 in the small bowel using VCE (video endoscopy); The Lewis score analyses 5 mucosal parameters for each of the four segments of the small bowel (duodenum, jejunum, proximal and distal ileum): erythema, oedema, presence of nodular lesions, ulcerations and stenosis. A Lewis score < 135 indicates inactive disease.
Proportion of endoscopic remissions according to the number of ulcerations | Week 24
  A patient is considered to be in endoscopic remission if they have:
  - no ulceration using endoscopic video capsule (VCE) at week 24;
Proportion of endoscopic remissions according to the Magnetic Resonance Imaging (MRI) activity | Week 24
  A patient is considered to be in endoscopic remission if they have:
  - no activity on MRI at week 24 (defined as segmental MaRIA score < 7); The MaRIA (Magnetic Resonance Index of Activity) scoring system is used to assess ileocolic Crohn's disease activity on contrast-enhanced MRI enterography. The segmental index represents the severity of disease in a segment of the bowel, while assessing six defined anatomical regions that can be combined to form an overall MaRIA index.
  The cut-off points for the MaRIA score are as follows:
  moderate disease: ≥7 severe disease: ≥11
Proportion of endoscopic remissions according to bowel thickness | Week 24
  A patient is considered to be in endoscopic remission if they have:
  - no bowel thickness on ultrasound at week 24 (< 3mm with no other signs of activity).
Treatment failure | Weeks : 24; 52
  Compare treatment failure at week 24 or week 52 in the 2 groups.
  Treatment failure is defined as:
  * The performance of a CD-related surgery between inclusion and week 24 ;
  * OR use of steroids between baseline and week 24;
  * OR treatment dose optimisation between inclusion and week 24;
  * OR a change in treatment between inclusion and week 24.
Adverse events | Week 24
  Compare the percentage of adverse events in both arms at week 52
Symptomatic remission at week 24 | Week 24
  Symptomatic remission at week 24 is a composite criterion measured by PRO2 defined as: Stool frequency (SF) < 3 with abdominal pain score (AP) < 2 at week 24; AND absence of therapeutic failure between inclusion and week 24.
Changes in quality of life score (Inflammatory Bowel Disease Questionnaire (IBDQ)-32 | Weeks : 0; 24
  Compare evolution of IBDQ-32 in the two groups of patients between inclusion and week 24.
  The IBDQ-32 questionnaire consists of 32 questions. Each question is answered on a scale from 1 to 7, with 1 being the lowest score and 7 the highest. Adding up the different scores gives a total score, ranging from 32 (worst score) to 224 (best score). The higher the score, the better the quality of life.
Clinical and biomarker remission | Weeks : 12; 52
  Compare rates of clinical and biomarker remission at week 12 and week 52.
Mucosal remission | Week 24
  Rate of Mucosal remission at week 24. Mucosal remission is definied by ;
  * a CDEIS score < 3 at week 24 using ileocolonoscopy ; The CDEIS is an index of the severity of intestinal lesions caused by Crohn's disease.
  * Or a Lewis score < 135 at week 24 in the small bowel using VCE (video endoscopy)
  * Or no ulceration using endoscopic video capsule (VCE) at week 24;
  * Or no activity on MRI at week 24 (defined as segmental MaRIA score < 7);
  * Or no bowel thickness on ultrasound at week 24 (< 3mm with no other signs of activity).
Clinical Decision Support Tool (CDST) score | Week 52
  Analyze the CDST score for prediction of remission under vedolizumab and adalimumab optimization.
  A CDST score :
  * < 13 points is considered a low probability of remission;
  * Between 13 and 19 points is considered an intermediate probability of remission;
  * > 19 points is considered a high probability of remission.

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde BARRAU, MD, Principal Investigator — CHU de Saint-Etienne
Locations (12):
- France (12):
  - APHP - Hôpital Bicêtre, Le Kremlin-Bicêtre, Paris
  - CHU Amiens, Amiens
  - CHRU Lille, Lille
  - Chu Limoges, Limoges
  - APHM, Marseille
  - CHU Montpellier, Montpellier
  - Hôpital de l'Archet II, Nice
  - Assistance Publique - Hôpitaux de Paris, Paris
  - CHU Bordeaux, Pessac
  - Ch Lyon Sud, Pierre-Bénite
  - CHU Rennes, Rennes
  - CHU de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No